CLINICAL TRIAL: NCT02744118
Title: Helping Eliminate Marijuana Use Through Pediatric Practice
Acronym: HEMPP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: American Academy of Pediatrics (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: AmericanAP; 5R21DA039326-02 (NIH)
Record Dates: First submitted 2016-03-30; First posted 2016-04-20 (Estimated); Last update posted 2020-07-09 (Actual); Status verified 2020-07

CONDITIONS: Marijuana
Keywords: Media Use
MeSH Terms: conditions — Marijuana Abuse

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Marijuana Screening and Brief Counseling (Experimental): The marijuana screening and brief counseling intervention will be developed based on a tested adolescent tobacco cessation intervention and the Public Health Service 5As model. The proposed intervention will be adapted using current literature, input from content experts, and qualitative data gathered using focus groups.
  Interventions: Other: 5A's Model
- Healthy Internet Use Model (Active Comparator): The media screening and brief counseling intervention is based on a media use screening and brief counseling intervention tested as the active comparator for a 5As tobacco cessation randomized control trial (NCT01312480) and the 2010 American Academy of Pediatrics policy statement on children and media.
  Interventions: Other: Healthy Internet Use Model

INTERVENTIONS:
Other: 5A's Model — The adapted 5A's model will include the following elements:
  1. Ask the patient about their marijuana use
  2. Advise every patient to quit/reduce marijuana use using clear, specific personalized advice
  3. Assess factors affecting choice of behavior and behavior change
  4. Assist abstinence/reduction in in marijuana use using behavior change techniques to aid the patient
  5. Arrange follow-up for ongoing assistance and support, and to adjust treatment plans
  Arms: Marijuana Screening and Brief Counseling
Other: Healthy Internet Use Model — The Healthy Internet Use Model provides a framework for conversations between pediatric practitioners and their adolescent patients. It focuses on 3 key areas of social media behavior:
  1. Balance
  2. Boundaries
  3. Communication
  Arms: Healthy Internet Use Model

SUMMARY:
This study adapts the Public Health Service (PHS) 5As model for use with adolescent marijuana users and pilot the intervention to test feasibility and acceptability in pediatric primary care settings. The specific aims are as follows:

Aim 1: Develop a marijuana screening and brief counseling intervention for adolescents based on the Public Health Service 5As model and previously developed adolescent smoking cessation intervention.

Hypothesis 1: The 5As model can be adapted for use as a marijuana screening and counseling intervention for adolescents.

Aim 2: Test the feasibility and acceptability of the 5As marijuana screening and brief counseling intervention in pediatric primary care practice.

Hypothesis 2a: Pediatric clinicians will find the 5As intervention feasible and acceptable for addressing marijuana use in routine clinical visits with adolescents and their families; and

Hypothesis 2b: Adolescents will find the 5As intervention delivered by their clinicians to be acceptable in the context of routine preventive services delivery.

DETAILED DESCRIPTION:
The HEMPP study involves three phases: Researchers will (1) Develop a marijuana screening and brief counseling intervention for adolescents, based on expert input, current literature, and themes gathered from focus groups with adolescents and clinicians; (2) Pilot test the acceptability of the 5As marijuana intervention in 2 pediatric primary care practices, where researchers will test the intervention and determine acceptability via in-depth interviews with clinicians, office staff, adolescents and parents; and (3) Pilot test the feasibility of the 5As marijuana intervention in 8 practices (4 intervention/4 comparable control), wherein each practice will enroll 100 adolescents and conduct baseline/exit interviews with all of them. Twenty percent of adolescents/practice (including identified marijuana users) will complete one follow-up interview 3-6 weeks after their practice visit. These interviews will assess physician-delivery of the intervention and any change in use, attitude or behavioral intentions toward marijuana since their clinical visit. Findings will inform the development of a future large-scale trial of adolescent marijuana use, screening and cessation counseling in pediatric primary care. The long-term goal is to improve clinical preventive services for adolescent marijuana cessation. Conducting this work within the AAP PROS network will lead to rapid dissemination of effective interventions.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents presenting for regular well or sick visits at their pediatrician's office
* Must live in a home or apartment with access to a telephone and mailing address
* Must be cognitively able to consider the risks of marijuana use
* Must be able to speak English
* Must be able and willing to give informed consent (if 18 years of age or older) or assent (if 14-17 years of age)
* In addition: parents/legal guardians of minors must be able and willing to give informed consent

Exclusion Criteria:

* None

Ages: 13 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 620 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2020-03 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
Change in Adolescent Marijuana Use and Habits at 3-6 Weeks using the Timeline Followback (TLFB) Method | Baseline (doctor's visit) and 3-6 weeks after doctor's visit
  Via a baseline survey and a phone interview 3-6 weeks later, using the Timeline Followback Method (TLFB), adolescents will be asked to report their current marijuana-use status, and will explore whether receiving the intervention affects motivation, intentions to quit and reduce use, or change in marijuana-use habits. Marijuana use will be defined as smoking or ingestion of any part of the marijuana plant; categories include: ever user, past month (current) user; past week and daily user. Addiction measures will include: compulsive use, psychoactive effects and drug-reinforced behaviors.

SECONDARY OUTCOMES:
Health and Behavioral Outcomes Related to Adolescent Marijuana Use | 3-6 weeks after initial doctor's visit
  Via a baseline survey and a phone interview 3-6 weeks later, using validated mental health and behavioral measures previously developed for longitudinal studies of neurodevelopmental impact of mercury exposure (Myers, 1995), modified for the current intervention. Specific outcomes include: cognitive and social functioning, psychomotor performance,health service utilization, development of dependence, school performance, and alcohol and other drug use. Changes in health and behaviors from before the clinical intervention will help determine short-term impact of the intervention on outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: V. Fan Tait, MD, Principal Investigator — American Academy of Pediatrics
Locations (1):
- American Academy of Pediatrics, Elk Grove Village, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2018-09-19): https://cdn.clinicaltrials.gov/large-docs/18/NCT02744118/ICF_000.pdf